CLINICAL TRIAL: NCT06408025
Title: Mental Health-App for Improving Depressive Symptoms
Brief Title: Syrenity App for Depression
Acronym: SYRA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Syra Health (Unknown)
Responsible Party: Principal Investigator, Lorenzo Lorenzo-Luaces, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22283; 2023-0410 (Other: Pearl IRB)
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Syrenity App (Experimental): The Syrenity App is a mental health app that has been designed to help improve mental health and well-being. The content on the app was created using cognitive-behavioral therapy principles. It uses both active and passive interventions. Active interventions are interventions where the user engages with the app in a back and forth dialogue (e.g., a conversation about restructuring unhelpful thoughts). Passive interventions meanwhile consist of text or videos that the user can read or watch and do not require dialogue with the app.
  Interventions: Other: Syrenity App
- Waiting list control (No Intervention): Those assigned to the waiting list control condition will complete weekly surveys as those assigned to the intervention group but will not have access to the Syrenity platform until after the the 6-week trial period.

INTERVENTIONS:
Other: Syrenity App — Currently, the Syrenity App has two active interventions. One is an exposure-based intervention called "Face your fears." Another is an intervention based on behavioral activation called "Get better." The app also provides self-report questionnaires for tracking mood along with psychoeducation on a variety of topics relevant to mental health.
  Arms: Syrenity App

SUMMARY:
The goal of this clinical trial is to learn if the Syrenity mental health app reduces depressive symptoms when compared to a control condition. Secondarily, the trial will provide data on the usability and acceptability of the Syrenity app. The main questions it aims to answer are:

Does Syrenity reduce self-reported depressive symptoms compared to a waiting list control? How usable is the Syrenity app?

ELIGIBILITY:
Inclusion Criteria:

* PHQ-9 >= 10
* Use an iPhone or Android
* Residing in the United States

Exclusion Criteria:

* PHQ-9 item 9 >= 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9 (PHQ-9) | 6 weeks
  Depression symptoms will be assessed with the PHQ-9. The PHQ-9 is a 9-item self-report measure that assesses the frequency of symptoms of major depressive disorder as outlined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-5). Response options range from 0 ("not at all") to 3 (nearly every day). Total scores on the PHQ-9 range from 0-27 with greater scores indicating greater frequency of depressive symptoms. A score greater than or equal to 10 on the PHQ-9 has been identified as a positive screen for major depression (Kroenke & Spitzer, 2002). PHQ-9 will be assessed at baseline, and each week of the intervention.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder Scale-7 (GAD-7) | 6 weeks
  Anxiety symptoms will be assessed with the GAD-7, a 7-item self-report measure that assesses the frequency of anxiety symptoms. Responses range from 0 ("not at all") to 3 ("nearly every day"), yielding total scores that range from 0-21 with greater scores indicating greater frequency of anxiety symptoms. A score greater than or equal to 10 on the GAD-7 has been identified as a positive screen for anxiety in primary care settings (Spitzer et al., 2006). GAD-7 will be assessed at baseline, and each week of the intervention.
Systems Usability Scale (SUS) | 6 weeks
  The SUS is a brief measure for assessing the usability of given systems (e.g., websites, mobile devices). The SUS has ten items and is rated on a five-point scale with responses ranging from zero ("strongly agree") to four ("strongly disagree"). Scale scores are multiplied by 2.5 to produce scores ranging from zero to 100 with higher scores indicating greater usability. We administered the SUS at the end of the intervention (week 6). However, investigators also administered a slightly modified version of the SUS at baseline to control for between-individual differences (e.g., the tendency to give high ratings). Participants were asked to rate their prediction of the usability of the book at baseline "based on the small amount of information [they] have on the study."

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No